CLINICAL TRIAL: NCT01716325
Title: E-support for Healthcare Processes - WEIGHT LOSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Primorska (Other)
Collaborators: National Institute of Public Health, Slovenia (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EHOW
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight loss - ICT support (Experimental): Weight loss - ICT support
  Interventions: Other: Self-management weight loss plan endorsement.
- Conventional (Other): Weight loss, comparator - no ICT support; conventional live workshops for weight loss
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Self-management weight loss plan endorsement. — Self-management weight loss plan endorsement.
  Arms: Weight loss - ICT support
Other: Conventional — Weight loss, comparator - no ICT support; conventional live workshops for weight loss
  Arms: Conventional

SUMMARY:
The purpose of the study is to establish and clinically evaluate a new approach to treating obesity by using information and communication technologies (ICT). A mobile environment and organizational interventions to improve the process of an integrated treatment of people with obesity will be identified, developed, introduced and clinically evaluated.

DETAILED DESCRIPTION:
A mobile environment to improve the process of an integrated treatment of obese people will be identified, developed, introduced and clinically evaluated. The study will include 150 patients aged between 25 to 65 for men and 25 to 70 for women, diagnosed with obesity (BMI≥30 or BMI>27,5 and 20% risk or more for developing a cardiovascular diseases). One group of patients will visit conventional live workshops for weight loss and the other group will use ICT. At the initial examination by the doctor all survey participants will have measured blood pressure, body mass, waist circumference, percentage of body fat, percentage of skeletal muscle, resting metabolic rate, estimated risk of developing cardiovascular disease and will be directed to laboratory examination (blood lipids and cholesterol, blood sugar). Both groups will go through 16 workshops for weight loss. Each week they will monitor their body mass, waist circumference, physical activity (type, duration, intensity) and food intake (type, quantity). After six months all survey participants will be examined again. We will compare effectiveness of ICT weight loss group with conventional weight loss group.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥30 or BMI>27,5 and 20% or more risk for developing a cardiovascular diseases
* Age between 25 - 65 years for men and 25 - 70 years for women
* Own a mobile phone
* Internet
* Know how to use a computer
* Know how to use an e-mail
* Signed voluntary consent to participate in the survey

Exclusion Criteria:

* People with movement disorders
* Age<18 years or age>70 years for women and 65 years for men
* Pregnancy, breast feeding, intention of getting pregnant during the study, period after childbirth (9 months)
* Does not own or know how to handle a mobile phone
* No internet access
* Known hospitalization for severe psychiatric disorders (schizophrenia, psychosis)
* Known history of eating disorders (anorexia, bulimia nervosa and others)
* Cancer incidence in the last 5 years
* Heart problems, chest pain, nausea, dizziness
* Chronic inflammatory diseases
* Other unregulated chronic diseases

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 16 weeks
  Weight loss of 5 to 10 % of the body mass at the beginning of the study

SECONDARY OUTCOMES:
Successful maintenance or improvement of the following measured parameter: Body mass index. | 16 weeks
Successful maintenance or improvement of the following measured parameter: waist circumference | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cirila Hlastan Ribič, PhD, Prof., Principal Investigator — National Institute of public Health
Locations (1):
- CINDI Slovenia, National Institute of Public Health, Ljubljana, Slovenia